CLINICAL TRIAL: NCT02780882
Title: A Proof of Concept and Open-label Study to Test the Efficacy and Safety of Pasireotide in Patients With Ectopic ACTH-producing Tumors
Brief Title: SOM230 Ectopic ACTH-producing Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to stringent inclusion/exclusion criteria, study investigator deemed it not feasible.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Ning-Ai Liu, MD, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro34493
Record Dates: First submitted 2016-04-26; First posted 2016-05-24 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Ectopic ACTH Syndrome
Keywords: Pasireotide; Ectopic ACTH; SOM230; ectopic ACTH-dependent Cushing's syndrome
MeSH Terms: conditions — ACTH Syndrome, Ectopic | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pasireotide (Experimental): Each patient will be treated with pasireotide at an initial dose of 600 μg twice daily for one month. The dose will be further increased to 900 μg twice daily for month 2 and 3. After month 3, patients who continue to meet the inclusion and exclusion criteria will be entered into an additional 3 months of treatment.
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Pasireotide
  Other Names: SOM230

SUMMARY:
The purpose of this prospective open-label phase II study, is to evaluate the efficacy of pasireotide twice daily subcutaneous injections for normalizing 24 hour urine free cortisol in patients with ectopic ACTH-producing tumors as measured by the proportion of patients achieving normal UFC at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any screening procedures
* Male or female patients aged 18 years or greater
* Confirmed non-pituitary ectopic-ACTH secreting tumor
* Well differentiated, and low or intermediate grade (WHO classification G1-2) neuroendocrine tumor
* Tumor size increase < 10% in 6 months prior to screening on CT or MRI
* Mean 24-hour urinary free cortisol level of at least 1.5 x the upper limit of the normal range, and a morning plasma ACTH level of > 5 ng/L

Exclusion Criteria:

* Patients with highly malignant ACTH-secreting tumors, i.e. small-cell lung carcinomas, medullary thyroid carcinomas, and pheochromocytomas
* Patients with poorly differentiated neuroendocrine tumors (WHO classification G3)
* Patients with >10% increase of tumor size in 6 months prior to screening by CT or MRI
* Patients with Cushing's syndrome due to pituitary ACTH secretion
* Patients with hypercortisolism secondary to adrenal tumors or nodular (primary) bilateral adrenal hyperplasia
* Patients who have a known inherited syndrome as the cause for hormone over secretion (i.e. Carney Complex, McCune-Albright syndrome, MEN-1)
* Patients with a diagnosis of glucocorticoid-remedial aldosteronism (GRA)
* Patients who have undergone major surgery within 1 month prior to screening
* Patients with known gallbladder or bile duct disease, acute or chronic pancreatitis (patients with asymptomatic cholelithiasis and asymptomatic bile duct dilation can be included)
* Diabetic patients whose blood glucose is poorly controlled as evidenced by HbA1C >8%
* Patients who have clinically significant impairment in cardiovascular function or are at risk thereof, as evidenced by
* Congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, clinically significant bradycardia, high grade AV block, history of acute MI less than one year prior to study entry
* QTcF >450 msec at screening

  * History of syncope or family history of idiopathic sudden death
  * Risk factors for Torsades de Pointes such as uncorrected hypokalemia, uncorrected hypomagnesemia, cardiac failure
  * Concomitant disease(s) that could prolong the QT interval such as autonomic neuropathy (caused by diabetes or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism, concomitant medication(s) known to increase the QT interval
* Patients with liver disease or history of liver disease such as cirrhosis, chronic active hepatitis B and C, or chronic persistent hepatitis, or patients with ALT or AST more than 2 x ULN, serum creatinine >2.0 x ULN, serum bilirubin >1.5 x ULN, serum albumin < 0.67 x LLN at screening
* Patients with any ongoing or planned anti-neoplastic therapy
* Has been treated with radionuclide at any time prior to study entry
* Is likely to require any additional concomitant treatment to pasireotide for the tumor
* Patients who have any current or prior medical condition that can interfere with the conduct of the study or the evaluation of its results, such as

  * History of immunocompromise, including a positive HIV test result (Elisa and Western blot). An HIV test will not be required, however, previous medical history will be reviewed
  * Presence of active or suspected acute or chronic uncontrolled infection
  * History of, or current alcohol misuse/abuse in the 12 month period prior to screening
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control. If a woman is participating in the trial then one form of contraception is sufficient (pill or diaphragm) and the partner should use a condom. If oral contraception is used in addition to condoms, the patient must have been practicing this method for at least two months prior to screening and must agree to continue the oral contraceptive throughout the course of the study and for 3 months after the study has ended. Male patients who are sexually active are required to use condoms during the study and for three month afterwards as a precautionary measure (available data do not suggest any increased reproductive risk with the study drugs)
* Patients who have participated in any clinical investigation with an investigational drug within 1 month prior to screening or patients who have previously been treated with pasireotide
* Known hypersensitivity to somatostatin analogues
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study
* Patients with presence of Hepatitis B surface antigen (HbsAg)
* Patients with presence of Hepatitis C antibody test (anti-HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of pasireotide twice daily subcutaneous injections for normalizing 24 hour urine free cortisol in patients with ectopic ACTH-producing tumors | 6 months
  Effectiveness of pasireotide as measured by 24 hour urine free cortisol

SECONDARY OUTCOMES:
Number of participants with abnormal laboratory values for urine free cortisol | 6 months
  Number of participants with abnormal laboratory values for hormones and metabolism as assessed by urine free cortisol
Number of participants with abnormal laboratory values for serum cortisol levels | 6 months
  Number of participants with abnormal laboratory values for hormones and metabolism as assessed by serum cortisol levels
Number of participants with abnormal laboratory values for salivary cortisol levels | 6 months
  Number of participants with abnormal laboratory values for hormones and metabolism as assessed by salivary cortisol levels
Number of participants with abnormal laboratory values for Hemoglobin A1C (HbA1C) | 6 months
  Number of participants with abnormal laboratory values for hormones and metabolism as assessed by Hemoglobin A1C (HbA1C)
Number of participants with abnormal laboratory values for fasting blood glucose | 6 months
  Number of participants with abnormal laboratory values for hormones and metabolism as assessed by fasting blood glucose
Number of participants with abnormal laboratory values for blood electrolytes | 6 months
  Number of participants with abnormal laboratory values for hormones and metabolism as assessed by blood electrolytes
Number of participants with abnormal laboratory values for plasma adrenocorticotropic hormone (ACTH) | 6 months
  Number of participants with abnormal laboratory values for hormones and metabolism as assessed by plasma adrenocorticotropic hormone (ACTH)
Number of participants with abnormal laboratory values for plasma beta-lipotropin | 6 months
  Number of participants with abnormal laboratory values for hormones and metabolism as assessed by plasma beta-lipotropin
Number of participants with changes in clinical signs and symptoms | 6 months
  Number of participants with changes in clinical signs and symptoms of Cushing's disease as defined by changes in weight, body mass index, and blood pressure
Changes in Tumor Size | From baseline at months 3 and 6
  To evaluate changes in tumor size
Number of participants with changes in blood chemistry (safety) | Baseline and 6 months
  Number of participants with abnormal laboratory values for blood chemistry as assessed by total proteins, amylase, lipase, total cholesterol (TC), low-density lipids (LDL)-cholesterol, m creatinine, creatinine clearance, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, albumin, alkaline phosphatase (ALP), gamma-glutamyl transferase (GGT)
Number of participants with changes in hematology (safety) | Baseline and 6 months
  Number of participants with abnormal laboratory values for hematology as assessed by prothrombin time (PT), and international normalized ratio (INR)
Number of participants with changes in cardiac activity | Baseline and 6 months
  Number of participants with changes in cardiac activity as measured by electrocardiogram (ECG)
Number of participants with changes in liver health | Baseline and 6 months
  Number of participants with changes in liver health as determined by an abdominal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ning-Ai Liu, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No